CLINICAL TRIAL: NCT01097200
Title: Anatomic and Functional Outcomes of Vaginal Mesh ( ELEVATE) Compared With Laparoscopic Sacrocolpopexy for Pelvic Organ Prolapse
Brief Title: Sacrocolpopexy Versus Vaginal Mesh Procedure for Pelvic Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Francisco Carmona (Other)
Collaborators: American Medical Systems (Industry)
Responsible Party: Sponsor-Investigator, Francisco Carmona, Chief of Department of OB GYN, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bataller01
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Vaginal Vault Prolapse; Enterocele; Uterine Prolapse; Cystocele; Rectocele
Keywords: sacrocolpopexy; meshes; sacrospinous ligament
MeSH Terms: conditions — Pelvic Organ Prolapse; Hernia; Uterine Prolapse; Cystocele; Rectocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elevate meshes (Other): The use of Elevate (American Systems trade mark) meshes for the treatment of pelvic prolapse.
  Interventions: Device: Elevate mesh
- Sacrocolpopexy (Other): Sacrocolpopexy for the correction of the prolapse
  Interventions: Device: Sacrocolpopexy

INTERVENTIONS:
Device: Elevate mesh — The correction of the prolapse can be made by this new technique.
  Other Names: Pelvic meshes
  Arms: Elevate meshes
Device: Sacrocolpopexy — Attach a mesh between the vagina and the promontorium.
  Other Names: Colpofixation
  Arms: Sacrocolpopexy

SUMMARY:
Pelvic prolapse is one of the most frequent pathology in Gynecology. Recurrency of the prolapse after primary surgery is relatively high, 15-30%. Sacrocolpopexy has showed to be effective but it requires a long learning curves and is more aggressive. New meshes techniques seem to be effective, as well, with less learning curve but they are expensive and there are no randomize studies published.

The investigators aim is to compare both techniques in terms of: anatomical and functional efficacy, cost, operating time and complications.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with one or more clinically significant anterior, apical, or posterior genital prolapse disorder(s)(symptomatic POP-Q stage II or higher) requiring surgical repair.

Exclusion Criteria:

* Investigator determines subject is not a candidate for surgical repair of her genital prolapse.
* Subject has had a prior prolapse procedure involving graft placement (synthetic or biologic)
* Subject has active or latent systemic infection or signs of tissue necrosis.
* Subject has restricted leg motion (inability to abduct or adduct leg positioning in the lithotomy position) with or without a hip replacement / prosthesis.
* Subject is currently pregnant or intends to become pregnant during the study period.
* Subject has had radiation therapy to the pelvic area.
* Subject has pelvic cancer, has had pelvic cancer within the past 12 months or has been on cytostatic medication within the past 12 months.
* Subject has uncontrolled diabetes.
* Subject is on any medication with could result in compromised immune response, such as immune modulators.
* Subject has undergone previous pelvic surgery < 6 months prior to enrollment in this study.
* Subject is unwilling or unable to give valid informed consent.
* Subject is unwilling or unable to comply with the requirements of the protocol, complete all quality of Life questionnaires and return for all follow-up visits.
* Subject with contraindications for laparoscopy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2016-11 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Functional and anatomical efficacy | 1 year

SECONDARY OUTCOMES:
operating time, cost and complications of both techniques | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bataller, M.D., Ph. D., Principal Investigator — Hospital Clinic, Barcelona, Spain.
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
First article has been submitted to the European Urology on feb 13th 2017, was rejected.
  Article accepted for publishing in may 2018 in IUJ

REFERENCES:
- [Background] Sanses TV, Shahryarinejad A, Molden S, Hoskey KA, Abbasy S, Patterson D, Saks EK, Weber LeBrun EE, Gamble TL, King VG, Nguyen AL, Abed H, Young SB; Fellows' Pelvic Research Network. Anatomic outcomes of vaginal mesh procedure (Prolift) compared with uterosacral ligament suspension and abdominal sacrocolpopexy for pelvic organ prolapse: a Fellows' Pelvic Research Network study. Am J Obstet Gynecol. 2009 Nov;201(5):519.e1-8. doi: 10.1016/j.ajog.2009.07.004. Epub 2009 Aug 28. PMID 19716533
- [Background] Cosson M, Rosenthal C, Clave H, et al. Prospective clinical assessment of the total transvaginal mesh (TVM) technique for treatment of pelvic organ prolapse-6 and 12 month results. Int Urogynecol J 2006; 17: S142.
- [Background] Nygaard IE, McCreery R, Brubaker L, Connolly A, Cundiff G, Weber AM, Zyczynski H; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy: a comprehensive review. Obstet Gynecol. 2004 Oct;104(4):805-23. doi: 10.1097/01.AOG.0000139514.90897.07. PMID 15458906